CLINICAL TRIAL: NCT02440958
Title: Modified FOLFIRINOX for Gemcitabine Refractory Pancreatic Cancer: A Phase II Multicenter Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0973
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- modified FOLFIRINOX (Experimental)
  Interventions: Drug: modified FOLFIRINOX regimen

INTERVENTIONS:
Drug: modified FOLFIRINOX regimen — Modified FOLFIRINOX regimen consisted of oxaliplatin at a dose of 60 mg per square meter, given as a 2-hour intravenous infusion, after 60 minutes, of irinotecan at a dose of 120 mg per square meter, given as a 90-minute intravenous infusion, immediately followed by leucovorin at a dose of 400 mg per square meter, given as a 2-hour intravenous infusion through a Y-connector. This treatment was immediately followed by fluorouracil at a dose of 400 mg per square meter, administered by intravenous bolus, followed by a continuous intravenous infusion of 2400 mg per square meter over a 46-hour period every 2 weeks

SUMMARY:
Pancreatic ductal adenocarcinoma is the fourth cause of death in the Western world. Surgery remains the only treatment offering an advantage in terms of overall survival (5-year survival range, 15-25%), but unfortunately only 10-20% of patients present resectable disease at the time of diagnosis. Since the approval of gemcitabine as a standard treatment for advanced pancreatic patients, no drug or combination of drugs has significantly improved the prognosis. Recently, as compared with gemcitabine, FOLFIRINOX was associated with a survival advantage (11.1 vs 6.8 months), but had increased toxicity. In some retrospective studies, modified FOLFIRINOX regimen (60/120 mg/m2 of oxaliplatin and irinotecan) has an improved safety profile in digestive malignancies. The purpose of this phase II multicenter study was to investigate the efficacy and safety in patients with pancreatic cancer who progressed in gemcitabine-based first line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed pancreatic ductal adenocarcinoma (metastatic or locally advanced stage)
* Refractory or progress to Gemcitabine based 1st line chemotherapy
* Older than 19 years old and younger than 75 years old
* Life expectancy> 3 months
* ECOG Performance status ≤2
* Only patients with measurable lesions in imaging study
* Adequete BM function (WBC ≥ 3,500/µl, absolute neutrophil cell count ≥ 1,500 /µl, platelet count ≥ 100,000/µl)
* Adequete liver function (total bilirubin < 1.5 X the upper limits of normal (ULN), AST and ALT <3 X UNL, and alkaline phosphatases < 3 X ULN or < 5 x ULN in case of liver involvement)
* Adequete renal function (serum creatinine < 1.5 mg/dl)
* Adequete cardiopulmonary function

Exclusion Criteria:

* Pathologically confirmed another type of pancreatic cancer (except ductal adenocarcinoma)
* Metastatic adenocarcinoma of originating at other organs
* Evidence with CNS metastasis
* Active infection
* Uncontrolled serious medical or psychiatric illness which can induce toxicity ro complication of treatment, such as inability to swallow, lacking physical integrity of the gastrointestinal tract, malabsorption syndrome, or active ulceration at upper gastrointestinal tract.
* Coexisting of other malignancies within 5 years, except squamous cell carcinoma and basal cell carcinoma of the skin
* Participation in any other investigational drug study within 1 month
* No signed informed consent

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08-28; Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
True response rate | within 16 weeks

SECONDARY OUTCOMES:
Overall survival | 6, 12 months